CLINICAL TRIAL: NCT01631981
Title: A Phase II, Multicentre, Randomised, Two-Arm, Parallel Group, Double-Blind, Placebo Controlled Study of the Steroid Sulfatase Inhibitor PGL2001 With Concomitant Administration of NETA (Norethisterone Acetate) for the Treatment of Symptoms Related to Endometriosis
Brief Title: PGL2001 Proof of Concept Study in Symptomatic Endometriosis
Acronym: AMBER
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: PregLem SA (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PGL11-007
Record Dates: First submitted 2012-06-19; First posted 2012-06-29 (Estimated); Last update posted 2014-06-03 (Estimated); Status verified 2014-06

CONDITIONS: Endometriosis
MeSH Terms: conditions — Endometriosis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- PGL2001 (Experimental): PGL2001 + NETA followed by NETA-only follow-up period
  Interventions: Drug: PGL2001 + Primolut-Nor 5
- Placebo (Placebo Comparator): Placebo + NETA followed by NETA-only follow-up period
  Interventions: Drug: Placebo + Primolut-Nor 5

INTERVENTIONS:
Drug: PGL2001 + Primolut-Nor 5 — PGL2001(estradiol sulfamate, E2MATE, ZK190628), Tablets, 1mg. 4 mg weekly for 4 weeks followed by 2mg weekly for 12 weeks.
  Norethisterone acetate (NETA), Tablets, 5mg. Once daily for 16 weeks plus during follow-up.
  Arms: PGL2001
Drug: Placebo + Primolut-Nor 5 — Placebo, Tablets.4 tablets weekly for 4 weeks followed by 2 tablets weekly for 12 weeks.
  Norethisterone acetate (NETA), Tablets, 5mg.Once daily for 16 weeks plus during follow-up.
  Arms: Placebo

SUMMARY:
This is a Phase II, multicentre, randomised, two-arm, parallel group ,double-blind, placebo controlled, study to investigate the efficacy, safety, pharmacokinetics and pharmacodynamics of the steroid sulfatase inhibitor PGL2001 with concomitant, continuous NETA administration for the treatment of pain symptoms suggestive of endometriosis. The target population will be women of reproductive age with symptoms suggestive of endometriosis.

ELIGIBILITY:
Inclusion Criteria:

* Provide written informed consent prior to initiation of any study related procedures.
* Be a woman of reproductive age between 18 and 45 years inclusive.
* Present with clinical signs suggestive of endometriosis.
* Be suffering from non menstrual pelvic pain and dysmenorrhea suggestive of endometriosis for at least 3 months prior to screening visit.

Exclusion Criteria:

* Be pregnant or currently lactating.
* Have diseases or suspected diseases which may cause pelvic pain not due to endometriosis.
* Have had any surgical treatment for endometriosis within the last 12 months.
* Have documented significant adenomyosis.
* Have participated in another clinical trial within the 30 days prior to the screening visit.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 162 (Actual)
Dates: Start 2012-06; Primary Completion 2013-10 (Actual); Study Completion 2014-05 (Actual)

PRIMARY OUTCOMES:
Non-menstrual pelvic pain. | Daily collection up to 16 weeks
  Use of a Visual Analogue Scale (VAS).

CONTACTS AND LOCATIONS:
Locations (20):
- Hungary (5):
  - Synexus Magyarország Kft., Budapest
  - Semmelweis Egyetem II. Szülészeti és Nőgyógyászati Klinika, Budapest
  - Debreceni Egyetem Orvos-es Egeszsegtudomanyi Centrum Szuleszeti es Nogyogyaszati Klinika, Debrecen
  - Pécsi Tudományegyetem Klinikai Központ Szülészeti és Nőgyógyászati Klinika, Pécs
  - Szegedi Tudományegyetem Szent-Györgyi Albert Klinkai Központ Szülészeti és Nőgyógyászati Klinika, Szeged
- Poland (10):
  - Medica Pro Familia Sp. z o.o. S.K.A. - Oddział Katowie, Katowice
  - Medeor Plus Szpital Wielospecjalistyczny, Lodz
  - Klinka Ginekologii Operacyjnej, Instytut-Centrum Zdrowia Matki Polki, Lodz
  - Specjalistyczny Gabinet Ginekologiczno-Położniczy, Lublin
  - Klinika Endokrynologii I Nieplodnosci Rozrodu, Ginekologiczno Polozniczy Szpital UM, Poznan
  - VitroLive Sp. Z o.o, Szczecin
  - Lubelskie Centrum Diagnostyczne, Świdnik
  - NZOZ Lecznica Medea, Warsaw
  - Private practice, Warsaw
  - Centralny Szpital Kliniczny MSWiA, Klinika Połoznictwa, Chorob Kobiecych i Ginekologii Onkologicznej, Warsaw
- Romania (5):
  - Euromedica Hospital SA, Baia Mare
  - Centrul Medical de Diagnostic si Tratament Ambulator Neomed SRL, Brasov
  - Genesys Fertility Center SRL, Bucharest
  - Centrul Medical Euromed SRL, Bucharest
  - Spitalul Clinic "Nicolae Malaxa", Bucharest